CLINICAL TRIAL: NCT06643780
Title: RANK-ligand Inhibition to Combat Sarcopenia with Underlying Osteoporosis: a Randomized, Double-blind, Double-dummy, Active-Controlled Trial
Brief Title: RANK-ligand Inhibition to Combat Sarcopenia with Underlying Osteoporosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ronald Man Yeung WONG, Clinical Associate Professor, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022.555
Record Dates: First submitted 2024-09-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Sarcopenia in Elderly
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Denosumab group (Active Comparator): 60mg subcutaneous Denosumab (1mL solution) every 6 months and intravenous placebo (100mL normal saline) once yearly
  Interventions: Drug: Denosumab
- Zolendronic acid group (Placebo Comparator): 5mg intravenous Zoledronic Acid (100mL solution) once yearly and subcutaneous placebo (1mL normal saline) every 6 months
  Interventions: Drug: Zolendronic Acid

INTERVENTIONS:
Drug: Denosumab — 60mg subcutaneous Denosumab (1mL solution) every 6 months and intravenous placebo (100mL normal saline) once yearly
  Arms: Denosumab group
Drug: Zolendronic Acid — 5mg intravenous Zoledronic Acid (100mL solution) once yearly and subcutaneous placebo (1mL normal saline) every 6 months
  Arms: Zolendronic acid group

SUMMARY:
The objective of this study was to conduct a randomized, double-blind, double-dummy active controlled trial to determine the efficacy of denosumab in treating sarcopenia with underlying osteoporosis.

DETAILED DESCRIPTION:
Aims:

1. To assess whether receptor activator of nuclear factor-kB ligand (RANKL)-inhibition can treat sarcopenia in osteosarcopenic patients, in terms of appendicular skeletal muscle mass (ASM), handgrip strength, and physical performance.
2. To assess whether RANKL-inhibition improves quality of life, and decreases falls, fractures, hospital admissions and mortality in osteosarcopenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Elderly males or females aged 65 years or older
* diagnosed with osteosarcopenia (sarcopenia diagnosis based on AWGS 2019 guidelines - low appendicular skeletal muscle mass (ASM) by Dual-energy X-ray absorptiometry (DXA) (M:<7.0kg/m2, F:<5.4kg/m2) AND low handgrip strength (M:<28kg, F:<18kg) OR low physical performance (6-metre walk: <1.0m/s or 5-time chair stand test ≥ 12 s); osteoporosis diagnosed based on World Health Organization (WHO) criteria with DXA scan T-score ≤ -2.5)
* Willing and able to comply with study protocol including follow-up evaluations.

Exclusion Criteria:

* history of recent fracture i.e., within 3 months
* history of prior anti-osteoporotic drug
* disease or medication affecting bone or muscle metabolism
* Chairbound or bedbound
* Unable to agree for consent
* contraindication to drug i.e., Denosumab or Zoledronic Acid
* Underlying malignancy or disease known to cause cachexia
* severe renal impairment e.g., Creatinine Clearance (CrCl) < 35ml/min
* moderate to severe liver failure (Child-Pugh Class B or C).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
6-metre walk | From enrollment to the end of treatment at 52 weeks
  The time taken to walk 6 metres without deceleration. Average result of 2 trials is recorded. Slow speed is defined as <1.0m/s.
5-time chair stand test | From enrollment to the end of treatment at 8 weeks
  The time to rise from a chair 5 times is recorded. The cut-off for is taken at >=12 seconds.
Appendicular skeletal muscle mass (ASM) | From enrollment to the end of treatment at 52 weeks
  Determined with Dual-energy X-ray absorptiometry (Horizon®, DXA system, Hologic, USA). Total ASM by DXA is evaluated by segmented measurement of muscle mass at four limbs by operator-defined cutlines at specific anatomical landmarks. ASM is adjusted to square of height to calculate ASMI (kg/m2). Low ASMI by DXA is < 7 kg/m2 for men and 5.4 kg/m2 for women.
Handgrip strength | From enrollment to the end of treatment at 52 weeks
  Assessed by spring-type hand dynamometer (JAMAR Hand Dynamometer 5030JO). Cut-off for men is < 28kg, and female is <18kg. Maximum reading of 3 trials using dominant hand in a maximum-effort isometric contraction
Quadriceps muscle strength | From enrollment to the end of treatment at 52 weeks
  Measured on affected limb with isometric dynamometer (Baseline, Genova, Italy). Subject will sit on a chair with both feet above ground, while raising the affected leg 45° forwards. The dynamometer is placed above the ankle and the subject will push the leg forward with maximum force. Measurements will be repeated 3 times and maximum value will be used for evaluation
Balancing ability | From enrollment to the end of treatment at 52 weeks
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes directional control (%).
Balancing ability | From enrollment to the end of treatment at 52 weeks
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes movement velocity (degrees/s)
Balancing ability | From enrollment to the end of treatment at 52 weeks
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes endpoint excursion (%)
Balancing ability | From enrollment to the end of treatment at 52 weeks
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes maximum excursion (%)
Balancing ability | From enrollment to the end of treatment at 52 weeks
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes reaction time(s)

SECONDARY OUTCOMES:
Falls | From enrollment to the end of treatment at 52 weeks
  To assess the occurrence of falls, patients are required to self-report via a fall calendar, which will be returned at 1-year
Fracture | From enrollment to the end of treatment at 52 weeks
  Assess occurrence of a fracture within a year of study period.
Quality of life Short Form-36 (SF-36) | From enrollment to the end of treatment at 52 weeks
  The highest score is 900, and the lowest score is 0. Highest score indicates a better quality of life.
Physical activity scale for elderly (PASE) | From enrollment to the end of treatment at 52 weeks
  It assesses the types of activities typically chosen by older adults, ranging from 0 to 793, with higher scores indicating greater physical activity
Food frequency questionnaire | From enrollment to the end of treatment at 52 weeks
  Daily and weekly intake of 280 food items will be performed using a validated food frequency questionnaire developed in a local population survey. Mean nutrient quantitation and energy intake per day will be calculated referring to food composition tables derived from the Chinese Medical Sciences Institute and Centre for Food Safety in Hong Kong.
Hospital admissions | From enrollment to the end of treatment at 52 weeks
  Number and cause of emergency hospital admission within 1 year of study period are documented.
Mortality | From enrollment to the end of treatment at 52 weeks
  Mortality within 1-year of study period is documented.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong RMY, Wong PY, Liu C, Tang N, Wan RCW, Liu WH, Cui C, Zhang N, Kwok TCY, Law SW, Cheung WH. RANK-ligand inhibition to combat sarcopenia with underlying osteoporosis: a study protocol for a randomized, double-blind, double-dummy, active-controlled trial. Trials. 2025 Aug 4;26(1):269. doi: 10.1186/s13063-025-08976-7. PMID 40760465